CLINICAL TRIAL: NCT01940380
Title: The Study of LTBP1 of Postmenopausal Women Osteoporosis Molecular Mechanism of Kidney Yang Deficiency Syndrome
Status: Completed | Type: Observational
Sponsor: Fujian Academy of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 20130305
Record Dates: First submitted 2013-09-04; First posted 2013-09-12 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Kidney Yang Deficiency Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Postmenopausal Osteoporosis is characterized by a decrease in bone mass as well as a deterioration of the bone architecture resulting in an increased risk of fracture,which is directly related to the lack of estrogen and also associated with a variety of genetic and acquired factors. Previous studies have found that POP molecular regulation mechanism of kidney Yang deficiency syndrome may be associated with LTBP1 gene expression.

This topic using RT-PCR and Western Blot detection POP of kidney Yang deficiency group and healthy group LTBP1 mRNA and proteion's expression level,validate LTBP1 relevance to POP the kidney Yang deficiency syndrome.To provide a scientific basis for clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

* • The Participants who volunteer to be test subjects, and can accept experimental drugs, and promise to finish the course should sign the informed consent.

  * Female ages 45 to 75 had gone through natural menopause before two years
  * In accordance with the western medicine diagnostic criteria of osteoporosis and belong to kidney Yin deficiency syndrome differentiation of traditional Chinese medicine certificate;
  * In accordance with the western medicine diagnostic criteria;
  * In accordance with TCM diagnostic methods; .If any of the above answers are no, The subjects couldn't in the study

Exclusion Criteria:

* Do not accord with standard of the western medicine diagnosis and TCM diagnostic methods

  * Age: <44 and > 76 years old;
  * With hyperparathyroidism, osteomalacia, rheumatoid arthritis, multiple myeloma and other serious complications such as secondary osteoporosis; Late or deformity, disability, loss of labor;
  * With cardiovascular, cerebrovascular, liver, kidney and hematopoietic system and other serious primary diseases;
  * Psychosis or alzheimer's patients;
  * Nearly three months, the use of hormone replacement therapy (HRT) and taking calcitonin, nearly six months has used double phosphonic acid salt for 15 days, etc.;
  * This medicine allergic constitution or composition of known to have allergies;
  * In a critical condition, It's difficult to make exact evaluators to efficacy and safety of the new drugs;

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female ages 45 to 75 had gone through natural menopause before two years
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2013-09 (Actual); Primary Completion 2013-12-01 (Actual); Study Completion 2016-12-09 (Actual)

PRIMARY OUTCOMES:
Postmenopausal Osteoporosis of kidney Yang deficiency syndrome | To observe the changes in gene expression(Day 1)

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Institute of Trational Chiness Medicine, Fuzhou, Fujian, China